CLINICAL TRIAL: NCT00747214
Title: A Multicenter, Randomized, Blinded Study Comparing the Effect of CRx-102 Plus DMARD Therapy to That of Placebo Plus DMARD Therapy on Serum C Reactive Protein (CRP) and Cytokines in Subjects With RA
Brief Title: A Study Comparing CRx-102 Plus Disease-modifying Anti-rheumatic Drug (DMARD) Therapy to Placebo Plus DMARD Therapy in RA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zalicus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRx-102-002
Record Dates: First submitted 2008-09-03; First posted 2008-09-05 (Estimated); Results first posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; RA; DMARD; CRP
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — dipyridamole, prednisolone drug combination; Prednisolone; Dipyridamole; Sugars

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRx-102 plus DMARD therapy (Experimental)
  Interventions: Drug: CRx-102; Drug: DMARD Therapy
- Placebo plus DMARD therapy (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: DMARD Therapy

INTERVENTIONS:
Drug: CRx-102
  Other Names: Prednisolone plus dipyridamole
  Arms: CRx-102 plus DMARD therapy
Drug: Placebo
  Other Names: sugar pill
  Arms: Placebo plus DMARD therapy
Drug: DMARD Therapy — DMARD therapy can include methotrexate or other DMARD therapy
  Other Names: Disease modifying anti-rheumatic drug therapy

SUMMARY:
This study was a Multicenter, Randomized, Blinded Study Comparing the Effect of CRx-102 Plus DMARD Therapy to that of Placebo Plus DMARD Therapy on Serum C Reactive Protein (CRP) and Cytokines in Subjects with Rheumatoid Arthritis. This Phase II, 6-week blinded study was planned for 60 subjects with moderate to severe rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
The primary objective of this study was to:

• Compare the response of CRx-102 plus DMARD therapy to placebo plus DMARD therapy in lowering CRP levels in rheumatoid arthritis subjects.

The secondary objectives of this study were to:

* Evaluate the changes in inflammatory cytokines in subjects treated with CRx-102 plus DMARD therapy to placebo plus DMARD therapy.
* Evaluate the efficacy of CRx-102 plus DMARD therapy to placebo plus DMARD therapy using ACR-20 and DAS28 indices as well as fatigue scales.

ELIGIBILITY:
Inclusion Criteria:

* Was 18 years of age of older
* Had moderate to severe RA
* Had at least 3 swollen joints (maximum 28) and 3 tender joints (maximum 28)
* Had a Baseline CRP level of at least 2.2 mg/L and a DAS28 score >4.5
* Had been on DMARD therapy for at least 3 months and have been on a stable dose of DMARD therapy for at least 28 days prior to enrollment
* Had a negative pregnancy test (females)
* Was not taking glucocorticoids at screening

Exclusion Criteria:

* Female subject is pregnant or lactating or of child bearing potential not using acceptable methods of birth control (barriers or abstinence). Female subjects using hormonal birth control are not to be enrolled.
* Subject is currently taking any steroids (glucocorticoids). All glucocorticoids must be discontinued for at least one month prior to entering study. Intraarticular, intramuscular, or intravenous glucocorticoids must not have been given at least 6 weeks prior to entering the study.
* Subject is currently taking more than 81 mg of aspirin daily.
* Subject is currently taking a statin, unless she/he has been on a stable dose of the same statin for at least 3 months prior to entering into the trial.
* Subject has any active infections or recent surgical procedures within 30 days of study initiation.
* Subject has uncontrolled diabetes mellitus as defined by a HbA1C value ≥ 7.0%.
* Subject knowingly has HIV or Hepatitis.
* Subject has undergone administration of any investigational drug within 30 days of study initiation.
* Subject has a history of hypersensitivity to steroids and/or dipyridamole.
* Subject has limited mental capacity or language skills such that simple instructions cannot be followed or information regarding adverse events cannot be provided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2004-11; Primary Completion 2006-09 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Lee, PhD, Study Director — Zalicus

RESULTS

PARTICIPANT FLOW:
Groups:
- CRx-102 Plus DMARD Therapy: Daily oral treatment with CRx-102, dosed twice per day (8AM and 1 PM) plus stable dose of DMARD therapy
  The following dose escalation scheme was used:
  Days 1 to 7 Dose level 1: CRx-102 (200 mg dipyridamole + 3 mg prednisolone)
  Days 8 to 42 Dose level 2: CRx-102 (400 mg dipyridamole + 3 mg prednisolone)
- Placebo Plus DMARD Therapy: Daily oral treatment with placebo, dosed twice per day (8AM and 1 PM) plus stable dose of DMARD therapy
Period: Overall Study
Arm/Group | CRx-102 Plus DMARD Therapy | Placebo Plus DMARD Therapy
Started | 27 | 32
Completed | 19 | 29
Not Completed | 8 | 3

BASELINE CHARACTERISTICS:
Population: Baseline analysis population is equal to the per protocol population defined as the subset of intent to treat population with no major protocol deviations including entry criteria and use of restricted medications and with study drug compliance of at least 75% during Days 1 to 42.
Groups:
- Total: Total of all reporting groups
Arm/Group | CRx-102 Plus DMARD Therapy | Placebo Plus DMARD Therapy | Total
Number analyzed (Participants) | 19 | 27 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (6.53) | 60.0 (12.25) | 58.5 (10.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 21 | 36
  Male | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in CRP From Baseline to Day 42
Description: The primary efficacy variable in this study was the change in CRP from Baseline (Day 1/Visit 2) to End of Study (Day 42/Visit 5). Blood samples for the analysis of serum CRP were taken at each visit.
Time Frame: Baseline and Day 42
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | CRx-102 Plus DMARD Therapy | Placebo Plus DMARD Therapy
Number analyzed (Participants) | 19 | 27
percentage change from baseline | -16.12 (94.99) | 9.60 (74.15)

2. Secondary Outcome: Improvement of ACR 20 Scores at End of Study (Day 42/Visit 5)
Description: The percentage of subjects in each group that achieved an ACR 20 response on Day 42
Time Frame: Day 42
Measure: Number; unit: percentage of participants
Arm/Group | CRx-102 Plus DMARD Therapy | Placebo Plus DMARD Therapy
Number analyzed (Participants) | 19 | 27
percentage of participants | 63 | 30

3. Secondary Outcome: Change in DAS28 Score From Baseline to Day 42
Description: To calculate the DAS28, the number of swollen joints and tender joints should be assessed using 28-joint counts, the ESR should have been measured in mm/hour, and the patient's general health (GH) or global disease activity measured on a Visual Analog Scale (VAS) of 100 mm must be obtained. Using these data, the DAS28 could be calculated using the following formula: DAS28 = 0.56 * sqrt(tender28) + 0.28 * sqrt(swollen28) + 0.70 * ln(ESR) + 0.014 * GH. The DAS28 provides a number between 0 and 10 that indicates the current activity of RA in the subject. A DAS28 above 5.1 means high disease activity and below 3.2 indicates low activity. Remission is achieved when a DAS28 score is lower than 2.6. The DAS28 measurements were to be taken at each visit.
Time Frame: Baseline and Day 42
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CRx-102 Plus DMARD Therapy | Placebo Plus DMARD Therapy
Number analyzed (Participants) | 19 | 27
units on a scale | -1.521 (1.574) | -0.697 (1.435)

4. Secondary Outcome: Change in Fatigue (MAF Scale) Score From Baseline to Day 42
Description: The Multidimensional Assessment of Fatigue (MAF) scale is a self-administered, 16 item questionnaire to measure self-reported fatigue (http://www.son.washington.edu/research/maf/). The following steps were used to calculate a single score ranging from 1 (no fatigue) to 50 (severe fatigue).
  1. Convert item #15 to a 0 to 10 scale by multiplying each score by 2.5
  2. Sum items #1, 2, and 3
  3. Average items #4 through 14
  4. Add results from above Steps 1 through 3 to obtain a single score
  A score was not be assigned to items #4 through 14 if a respondent indicated they "did not engage any activity for reasons other than fatigue." If respondent selected "no fatigue" on item #1, a 0 was to be assigned to items #2 through 16; item #16 was not included in the global fatigue index.
Time Frame: Baseline and Day 42
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CRx-102 Plus DMARD Therapy | Placebo Plus DMARD Therapy
Number analyzed (Participants) | 19 | 27
units on a scale | -7.840 (10.605) | -2.965 (9.186)

ADVERSE EVENTS:
Time Frame: 8 weeks: from screening (visit 1) up to 14 days prior to baseline (visit 2) through end of study (visit 5) on day 42.
Groups:
- CRx-102 Plus DMARD Therapy: Daily oral treatment with CRx-102, dosed twice per day (8AM and 1 PM) plus stable dose of DMARD therapy
  The following dose escalation scheme was used:
  Days 1 to 7 Dose level 1: CRx-102 (200 mg dipyridamole + 3 mg prednisolone) or placebo equivalent Days 8 to 42 Dose level 2: CRx-102 (400 mg dipyridamole + 3 mg prednisolone) or placebo equivalent
Arm/Group | CRx-102 Plus DMARD Therapy | Placebo Plus DMARD Therapy
Serious Adverse Events (participants affected / at risk) | 0/27 | 1/32
Other Adverse Events (participants affected / at risk) | 20/27 | 13/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRx-102 Plus DMARD Therapy (N=27) | Placebo Plus DMARD Therapy (N=32)
femoral hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) — Left femoral hernia that required hospitalization and surgical correction. In the opinion of the investigator this event was not related to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CRx-102 Plus DMARD Therapy (N=27) | Placebo Plus DMARD Therapy (N=32)
Headache (Nervous system disorders) | 13 | 0
Nausea (Gastrointestinal disorders) | 7 | 2
Vomiting (Gastrointestinal disorders) | 6 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 5
Dizziness (Nervous system disorders) | 3 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less